CLINICAL TRIAL: NCT03156504
Title: The BIO-K Study: A Single-Arm, Open-Label, Biomarker Development Clinical Trial of Ketamine for Non-Psychotic Unipolar Major Depression and Bipolar I or II Depression.
Acronym: Bio-K
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Network of Depression Centers (Other)
Responsible Party: Principal Investigator, Jennifer L. Vande Voort, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16-009737
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Results first posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Major Depression; Bipolar I Disorder; Bipolar II Disorder; Unipolar Depression
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Depressive Disorder | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketamine (Experimental): Subjects will receive three IV Ketamine Hydrochloride infusions (0.5 mg/kg, infused over 100 minutes) and measure their depressive symptom responses. Biomarkers will be developed using blood samples from study subjects, taken prior to (predictive biomarkers) and following ketamine treatment (change biomarkers).
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Subjects will receive three IV ketamine infusions at 0.5 mg/kg, infused over 100 minutes.
  Other Names: Ketalar

SUMMARY:
The purpose of this research study is to find out if the medication known as ketamine can help the symptoms of depression. This drug is approved by the Food and Drug Administration (FDA) but the investigators will use it for a non-FDA approved reason (depression).

DETAILED DESCRIPTION:
The investigators will enroll 100 adults with treatment-resistant unipolar or bipolar major depression (TRD) across 7 clinical sites and provide three IV ketamine infusions (0.5 mg/kg, infused over 100 minutes) and measure their depressive symptom responses. Biomarkers will be developed using blood samples from study subjects, taken prior to (predictive biomarkers) and following ketamine treatment (change biomarkers). The investigators will begin by studying the predictive value of mechanistic target of rapamycin (mTOR) target engagement by ketamine using a white blood cell (WBC) assay for antidepressive response to ketamine (Aim 1); however, samples will be used to develop multiple blood-based biomarkers for ketamine antidepressive effects (Aim 2). The investigators will also examine the effect of combining multiple blood-based biomarkers for predicting antidepressive response to ketamine in adults with TRD (Aim 3).

Baseline WBC markers of impaired cellular energy regulation will be associated with measures of clinical response to ketamine (predictive biomarker). Changes in WBC markers of impaired cellular energy regulation will be associated with clinical response to ketamine (change biomarker).

ELIGIBILITY:
Inclusion criteria:

* Ability to provide informed consent
* Current psychiatric inpatient (voluntary only) or outpatient treatment
* Meets Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnostic criteria for major depressive disorder, bipolar I disorder, or bipolar II disorder
* Patient Health Questionnaire (PHQ-9) total score > 15 at screening and at baseline (just prior to first acute phase ketamine infusion);
* Treatment-resistant depression, as defined by failure of at least two previous antidepressant or mood stabilizing treatments within the current depressive episode
* Failed antidepressant or mood stabilizing treatments can include pharmacotherapy for depression at an adequate dose for at least 8 weeks, or an acute series of at least 6 administrations of electroconvulsive therapy (ECT)
* Ability to pass a comprehension assessment test related to effects of ketamine and trial objectives and criteria

Exclusion Criteria:

* Diagnosis of schizophrenia, schizoaffective disorder, or active psychotic symptoms
* Ongoing prescription of > 4 mg lorazepam equivalents (total) daily, or morning dosing of any benzodiazepine at the time of assessment
* Currently undergoing ECT, transcranial magnetic stimulation, vagal nerve stimulation, or deep brain stimulation as either an acute or maintenance treatment of depression
* Any active or unstable medical condition judged by the study psychiatrist as conferring too great a level of medical risk to allow inclusion in the study
* Use or abuse of methamphetamine, cocaine, cannabis, or stimulants (prescribed and illicit) within the past 12 months
* Any current abuse or dependence of alcohol or drugs (excluding nicotine and caffeine) Note: Persons will be allowed to enroll in this study if their drug or alcohol abuse/dependence is in complete (not partial) and sustained (> 1 year) remission
* History of traumatic brain injury that resulted in loss of consciousness
* Developmental delay, mental retardation, or intellectual disorder
* Clinical or self-reported diagnosis of delirium, encephalopathy, or related clinical diagnosis within the prior 12 months
* Cognitive disorder (mild and major categories, per DSM-5)
* Prior participation in another study of ketamine for depression within the prior 6 months
* History of either poor antidepressive response to or poor tolerability of ketamine (any route of administration) when previously administered for treating symptoms of depression
* History of hypothyroidism unless taking a stable dose of thyroid medication and asymptomatic for 6 months
* Significant unstable medical condition
* Hepatic insufficiency (2.5 X upper limit of normal (ULN) for aspartate aminotransferase (AST) or ALT) within 1 year of consent, past liver transplant recipient, and/or clinical diagnosis of cirrhosis of the liver
* Pregnancy, or nursing
* Prisoners
* Involuntary psychiatric hospitalization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Frye, MD, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Cincinnati Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh B, Parikh SV, Voort JLV, Pazdernik VK, Achtyes ED, Goes FS, Yocum AK, Nykamp L, Becerra A, Smart L, Greden JF, Bobo WV, Frye MA, Burdick KE, Ryan KA. Change in neurocognitive functioning in patients with treatment-resistant depression with serial intravenous ketamine infusions: The Bio-K multicenter trial. Psychiatry Res. 2024 May;335:115829. doi: 10.1016/j.psychres.2024.115829. Epub 2024 Feb 28. PMID 38479192
- [Derived] Parikh SV, Vande Voort JL, Yocum AK, Achtyes E, Goes FS, Nykamp L, Singh B, Lopez-Vives D, Sera CE, Maixner D, Tarnal V, Severe J, Bartek S, Tye SJ, Rico J, Stoppel CJ, Becerra A, Smart L, Miller CR, Frye MA, Greden JF, Bobo WV. Clinical outcomes in the biomarkers of ketamine (Bio-K) study of open-label IV ketamine for refractory depression. J Affect Disord. 2024 Mar 1;348:143-151. doi: 10.1016/j.jad.2023.12.033. Epub 2023 Dec 22. PMID 38142892
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine
Started | 75
Completed | 74
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ketamine
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.27 (12.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 73
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 72
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 75

OUTCOME MEASURES:

1. Primary Outcome: Clinical Remission of Depression
Description: Total number of subjects with ≤ 9 MADRS score 24 hours post Ketamine infusion #3. The Montgomery Åsberg Depression Scale (MÅDRS) is a 10-item observer rating scale assessing symptoms of depression. The score ranges from 0 (no depression) to 60 (very depressed). For this study a score of less than or equal to 9 was considered clinical remission of depression.
Time Frame: 24 hours post infusion #3
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine
Number analyzed (Participants) | 74
Participants | 39

2. Primary Outcome: Suicidal Ideation
Description: Total number of subjects to have a reduction of suicidality, as defined by a 50% reduction on the Beck Scale for Suicidal Ideation (BSS) 24 hours post Ketamine infusion #3. The Beck Scale for Suicidal Ideation consists of 19 items which can be used to evaluate a patient's suicidal intentions. Each of the 19 items is rated on a 0-3 point scale (range 0-38, with higher scores indicating greater suicidal ideations or risk), and includes specific items that assess wish to live, wish to die, desire to make an active suicide attempt, passive suicidal desire, duration of suicidal ideations, frequency of suicidal ideations, and subjective level of control over suicidal actions.
Time Frame: 24 hours post infusion #3
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine
Number analyzed (Participants) | 74
Participants | 42

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately 5-7 weeks on all participants
Arm/Group | Ketamine
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 3/75
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=75)
Lightheadedness with low blood pressure (General disorders) | 1 (1)
Pump Malfunction (Product Issues) | 1 (1)
PTSD (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT03156504/Prot_SAP_000.pdf